CLINICAL TRIAL: NCT03021902
Title: Nutrition and Exercise in Critical Illness (The NEXIS Trial): A Randomized Trial of Combined Cycle Ergometry and Amino Acids in the ICU
Brief Title: Nutrition and Exercise in Critical Illness
Acronym: NEXIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clinical Evaluation Research Unit at Kingston General Hospital (Other)
Collaborators: University of Vermont (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Daren K. Heyland, Director, Clinical Evaluation Research Unit at Kingston General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: The NEXIS Trial
Record Dates: First submitted 2016-12-21; First posted 2017-01-16 (Estimated); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Acute Respiratory Failure
MeSH Terms: interventions — Amino Acids; Injections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- IV amino acid + in-bed cycle ergometry (Experimental): Beginning within 96 hours of initiation of mechanical ventilation, participants will receive the combined intervention that includes IV amino acids supplementation and in-bed cycle ergometry exercise
  Interventions: Drug: IV amino acids; Device: In-bed cycle ergometry exercise
- Usual care (No Intervention): Participants randomized to the usual care arm will receive usual care protein and exercise.

INTERVENTIONS:
Drug: IV amino acids — IV amino acids delivered by continuous infusion, such that the total enteral and IV protein will be between 2.0-2.5 g/kg/day as a combination of amino acid infusion plus standard feeding.
  Other Names: Clinisol 15% (Baxter) - sulfite-free (Amino Acid) Injection
  Arms: IV amino acid + in-bed cycle ergometry
Device: In-bed cycle ergometry exercise — In-bed cycle ergometry exercise delivered in 45-minute sessions once-daily 5 days per week according to a detailed specific protocol that includes a safety check in combination with vigorous verbal encouragement from trained research staff delivering the intervention to promote active cycling.
  Cycling is protocolized to provide graduated increases in resistance during each session and between daily sessions. Cycling will continue through ICU discharge or 21 calendar days after randomization. The intervention will specifically occur during ICU stay.
  Other Names: MotoMed Letto II Cycle Ergometer
  Arms: IV amino acid + in-bed cycle ergometry

SUMMARY:
This study proposes a novel early intervention combining Intravenous (IV) amino acids plus in-bed cycle ergometry exercise to improve physical outcomes in critically ill patients. The investigators hypothesize that this innovative approach will improve short-term physical functioning outcomes (primary outcome), as well as amino acid metabolism, body composition, and patient-reported outcomes at 6-month follow-up.

DETAILED DESCRIPTION:
The evaluation of a combination of exercise and protein supplementation in intensive care unit (ICU) patients is novel and potentially very important. For instance, outside of the ICU, in other clinical conditions, the combination of protein supplementation and exercise improves protein synthesis, muscle mass, and muscle strength compared to protein or exercise alone.[63-70] Hence, an opportunity exists to improve ICU patients' physical outcomes via evaluating the combination of optimized protein intake and early exercise in the ICU setting.

The proposed intervention and hypothesis: The investigators propose a multi-centered Phase II RCT, with blinded outcomes assessment, of a combination of intravenous (IV) amino acid supplementation and early in-bed cycle ergometry exercise versus usual care in ICU patients requiring mechanical ventilation. The investigators hypothesize that this novel combined intervention will: (1) improve physical functioning at hospital discharge; (2) reduce muscle wasting with improved amino acid metabolism and protein synthesis in-hospital; and (3) improve health-related quality of life, physical functioning, and healthcare resource utilization at 6 months after enrollment. Preliminary data show feasibility and safety of IV amino acids and the proposed exercise intervention. The investigators have chosen a primary outcome that correlates well with long-term outcomes including mortality, hospitalization, and quality of life. [54] If this Phase II trial is positive, investigators will seek funding for a Phase III RCT to demonstrate sustained improvements with a longer-term patient-centered primary outcome and to examine the feasibility, and facilitators/barriers of delivery of this intervention by ICU nurses, physical therapists, and others. If proven effective, this combined intervention has potential to revolutionize care of ICU patients and have a major public health impact on the growing number of ICU survivors.

Objectives: To demonstrate that the innovative combination of amino acid supplementation plus early in-bed cycle ergometry exercise improves physical outcomes of ICU patients.

Specific Aims of Full Phase II RCT:

1. Short-term performance-based physical function outcomes. To determine if a combined IV amino acid supplementation and in-bed cycle ergometry exercise intervention, compared to usual care, improves in hospital muscle strength and performance-based physical functioning outcomes in critically ill patients, using a primary endpoint of six-minute walk distance (6MWD) at hospital discharge.
2. Body composition. To determine if the combined intervention, compared to usual care, improves amino acid utilization and decreases muscle wasting in ICU patients (secondary endpoints).
3. Patient-reported outcomes and health care utilization at 6 months. To determine if the combined intervention, compared to usual care, improves physical functioning, health-related quality of life, and healthcare utilization at 6 months after study enrollment (secondary endpoints).

NEXIS Flame mechanisitic Ancillary sub study:

In the proposed sub-study, the addition of bronchoaveloar lavages, blood sampling and muscle sampling measures during the participant's ICU stay will provide the ability to examine the effects of the NEXIS intervention on inflammation as a possible mechanism for improved muscle weakness.

Specific Aims of the NEXIS FLAME mechanistic ancillary study:

1. To determine if the NEXIS intervention attenuates the release of IL-17 and related cytokines to reduce systemic inflammation in humans.
2. To determine if the NEXIS intervention reduces lung injury and neutrophilic lung inflammation in humans.
3. To determine if the NEXIS intervention attenuates skeletal muscle fiber atrophy via down regulation of muscle proteolytic pathways.
4. To determine if the NEXIS intervention, and exercise specifically, reduces the content of inflammatory cells in skeletal muscle.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old.
2. Requiring mechanical ventilation with actual or expected total duration of mechanical ventilation ≥ 48 hours.
3. Expected ICU stay ≥ 4 days after enrollment (to permit adequate exposure to the proposed intervention).

Exclusion Criteria:

1. >96 continuous hours of mechanical ventilation before enrollment.
2. Expected death or withdrawal of life-sustaining treatments within this hospitalization.
3. No expectation for any nutritional intake within the subsequent 72 hours.
4. Severe chronic liver disease (MELD score ≥20) or acute fulminant hepatitis.
5. Documented allergy to the amino acid intervention.
6. Metabolic disorders involving impaired nitrogen utilization
7. Not ambulating independently prior to illness that lead to ICU admission (use of gait aid permitted).
8. Pre-existing primary systemic neuromuscular disease (e.g. Guillain Barre).
9. Neuromuscular blocker infusion (eligible once infusion discontinued if other inclusion criteria met).
10. Intracranial or spinal process affecting motor function
11. Pre-existing cognitive impairment or language barrier that prohibits outcomes assessment.
12. Patients in hospital >5 days prior to ICU admission
13. Lower extremity impairments that prevent cycling (e.g. amputation, knee/hip injury).
14. Remaining intubated for airway protection only
15. Weight ≥150kg
16. Physician declines patient enrollment
17. Insufficient IV access
18. Pregnant
19. Incarcerated
20. Patients with acute kidney injury (AKI) as defined by meeting any of the KDIGO criteria (below) and not receiving renal replacement therapy:

    1. Increase in serum creatinine by ≥ 0.3 mg/dl within 48 hours or
    2. Increase in serum creatinine to ≥ 1.5 times baseline** or
    3. Urine volume <0.5 ml/kg/h for 6 hoursⴕ

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2025-01-14 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
Physical functioning | Hospital discharge (up to 26 weeks after randomization)
  6-minute walk distance

SECONDARY OUTCOMES:
Overall strength-upper extremity | Hospital discharge (up to 26 weeks after randomization)
  MRC Sum-score (Medical Research Council (MRC) Scale for Muscle Strength). Subscales scored 0-5, where 5 is normal. Total score is the sum of the 6 upper extremity subscales.
Overall strength-lower extremity | Hospital discharge (up to 26 weeks after randomization)
  MRC Sum-score (Medical Research Council (MRC) Scale for Muscle Strength). Subscales scored 0-5, where 5 is normal. Total score is the sum of the 6 lower extremity subscales.
Quadriceps force-lower extremity strength | Hospital discharge (up to 26 weeks after randomization)
  Hand held dynamometry
Distal strength-hand grip strength | ICU and hospital discharge (up to 26 weeks after randomization)
  Hand held dynamometry
Overall Physical Functional status - Short Physical Performance Battery | ICU and hospital discharge (up to 26 weeks after randomization)
  Short Physical Performance Battery
Overall Physical Functional status - Functional Status Score - ICU | ICU and hospital discharge (up to 26 weeks after randomization)
  Functional Status Score - ICU 5 items are performed: rolling, transfer from supine to sit, sitting at the edge of bed, transfer from sit to stand, and walking Each task is evaluated using an eight-point ordinal scale ranging from 0 (unable to perform) to 7 (complete independence) Item scores are summed The total score ranges from 0-35, with higher scores indicating better physical functioning.
Mortality | ICU and hospital discharge (up to 26 weeks after randomization)
  Chart review
Length of ventilation | ICU and hospital discharge (up to 26 weeks after randomization)
  Chart review
ICU stay | ICU and hospital discharge (up to 26 weeks after randomization)
  Chart review
Hospital stay | ICU and hospital discharge (up to 26 weeks after randomization)
  Chart review
ICU readmission | Hospital discharge (up to 26 weeks after randomization)
  Chart review
Re-intubation | Hospital discharge (up to 26 weeks after randomization)
  Chart review
Hospital-acquired infections | Hospital discharge (up to 26 weeks after randomization)
  Chart review
Discharge location (e.g. home vs. rehab) | Hospital discharge (up to 26 weeks after randomization)
  Chart review
Body composition - Ultrasound | Enrollment, hospital discharge, & ICU discharge (up to 26 weeks after randomization)
  Ultrasound of quadriceps
Body composition - CT - Chest when clinically available | Enrollment, hospital discharge, & ICU discharge (up to 26 weeks after randomization)
  Chest CT
Body composition - CT - Abdominal Scan when clinically available | Enrollment, hospital discharge, & ICU discharge (up to 26 weeks after randomization)
  Abdominal CT scan at 3rd lumbar vertebra
Health-related quality of life - SF-36 | Telephone survey at 6 months
  36-Item Short Form Health Survey (SF-36) All items are scored so that a high score defines a more favorable health state.
  Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100 Items in the same scale are averaged together to create the 8 scale scores. Items that are left blank (missing data) are not taken into account when calculating the scale scores.
  Scale scores represent the average for all items in the scale that the respondent answered.
Health-related quality of life - EQ-5D-5L | Telephone survey at 6 months
  EuroQol Group standardized measure of health status (EQ-5D-5L)
Physical functioning - Katz ADL | Hospital discharge (proxy) and telephone survey at 6 months
  Katz Index of Independence in Activities of Daily Living (Katz ADL) Total score where 6 = High (patient independent) 0 = Low (patient very dependent)
Physical functioning - Lawton IADL | Telephone survey at 6 months
  Lawton Instrument Activities of Daily Living Scale (Lawton IADL) A summary score ranges from 0 (low function, dependent) to 8 (high function, independent) for women and 0 through 5 for men to avoid potential gender bias.
Physical functioning/participation - return to work | Telephone survey at 6 months
  Return to baseline work/activity
Physical functioning/participation - living location | Telephone survey at 6 months
  Living location
Mental and Cognitive Functioning - MoCA-BLIND | Telephone survey at 6 months
  MoCA-BLIND The total possible score is 22 points; a score of 18 or above is considered normal
Mental and Cognitive Functioning - HADS | Telephone survey at 6 months
  Hospital Anxiety and Depression Scale The HADS questionnaire has seven items each for depression and anxiety subscales. Scoring for each item ranges from zero to three, with three denoting highest anxiety or depression level. A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depression.
Mental and Cognitive Functioning - IES-R | Telephone survey at 6 months
  Impact of Events Scale Scoring for each item ranges from 0-4 Total score ranges from 0-88, where a total score of 33 or over signifies the likely presence of PTSD
Health Care Resource Utilization | Telephone survey at 6 months
  Admission to ICU, hospital, rehabilitation & nursing facility
Body composition - DEXA Scan | At Hospital Discharge
  Whole Body DEXA Scan
Body Composition - Heavy water | Enrollment, Days 1-7
  Fat-free and fat mass can be measured with D2O in body fluids using gas chromatography-tandem mass spectrometry.
Plasma and muscle protein synthesis - Heavy water | Enrollment, Days 1-7
  Muscle protein synthesis will be analyzed with chromatography and mass spectrometry techniques.
NEXIS FLAME - Circulating inflammatory mediators | Enrollment, Days 3, 5, and 8
  Blood IL-17, IL-23, IL-6, TNFα, CXCK1, CXCL5, CXCL8, CCL2, SP-D, KL-6, vWF, and leukocyte counts with differential
NEXIS FLAME - Lung Inflammation | Enrollment, Day 5
  Bronchoalveolar lavage neutrophil counts, IL-17A, CXCL5, and protein
NEXIS FLAME - Muscle area | Enrollment, Day 5
  Single muscle fiber cross-sectional area (CSA), UPS expression, MuRF1 expression, myosin protein content (all from vastus lateralis sampling)
NEXIS FLAME - Muscle inflammation | Enrollment, Day 5
  Muscle macrophages (CD45+, CD206+)

CONTACTS AND LOCATIONS:
Overall Officials: Daren K Heyland, MD, MSc, Principal Investigator — Queen's University; Renee D Stapleton, MD, PhD, Principal Investigator — University of Vermont; Dale M Needham, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (7):
- United States (7):
  - University of Kentucky, Lexington, Kentucky
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Montefiore Albert Einstein College of Medicine, The Bronx, New York
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - University of Vermont College of Medicine, Burlington, Vermont
  - Harborview Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.

REFERENCES:
- [Background] Burtin C, Clerckx B, Robbeets C, Ferdinande P, Langer D, Troosters T, Hermans G, Decramer M, Gosselink R. Early exercise in critically ill patients enhances short-term functional recovery. Crit Care Med. 2009 Sep;37(9):2499-505. doi: 10.1097/CCM.0b013e3181a38937. PMID 19623052
- [Background] Chan KS, Pfoh ER, Denehy L, Elliott D, Holland AE, Dinglas VD, Needham DM. Construct validity and minimal important difference of 6-minute walk distance in survivors of acute respiratory failure. Chest. 2015 May;147(5):1316-1326. doi: 10.1378/chest.14-1808. PMID 25742048
- [Background] Kho ME, Truong AD, Zanni JM, Ciesla ND, Brower RG, Palmer JB, Needham DM. Neuromuscular electrical stimulation in mechanically ventilated patients: a randomized, sham-controlled pilot trial with blinded outcome assessment. J Crit Care. 2015 Feb;30(1):32-9. doi: 10.1016/j.jcrc.2014.09.014. Epub 2014 Sep 22. PMID 25307979
- [Background] Heyland D, Muscedere J, Wischmeyer PE, Cook D, Jones G, Albert M, Elke G, Berger MM, Day AG; Canadian Critical Care Trials Group. A randomized trial of glutamine and antioxidants in critically ill patients. N Engl J Med. 2013 Apr 18;368(16):1489-97. doi: 10.1056/NEJMoa1212722. PMID 23594003
- [Background] National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network; Rice TW, Wheeler AP, Thompson BT, Steingrub J, Hite RD, Moss M, Morris A, Dong N, Rock P. Initial trophic vs full enteral feeding in patients with acute lung injury: the EDEN randomized trial. JAMA. 2012 Feb 22;307(8):795-803. doi: 10.1001/jama.2012.137. Epub 2012 Feb 5. PMID 22307571
- [Background] National Heart, Lung, and Blood Institute ARDS Clinical Trials Network; Truwit JD, Bernard GR, Steingrub J, Matthay MA, Liu KD, Albertson TE, Brower RG, Shanholtz C, Rock P, Douglas IS, deBoisblanc BP, Hough CL, Hite RD, Thompson BT. Rosuvastatin for sepsis-associated acute respiratory distress syndrome. N Engl J Med. 2014 Jun 5;370(23):2191-200. doi: 10.1056/NEJMoa1401520. Epub 2014 May 18. PMID 24835849
- [Background] Parry SM, Berney S, Koopman R, Bryant A, El-Ansary D, Puthucheary Z, Hart N, Warrillow S, Denehy L. Early rehabilitation in critical care (eRiCC): functional electrical stimulation with cycling protocol for a randomised controlled trial. BMJ Open. 2012 Sep 13;2(5):e001891. doi: 10.1136/bmjopen-2012-001891. Print 2012. PMID 22983782
- [Background] Fan E, Zanni JM, Dennison CR, Lepre SJ, Needham DM. Critical illness neuromyopathy and muscle weakness in patients in the intensive care unit. AACN Adv Crit Care. 2009 Jul-Sep;20(3):243-53. doi: 10.1097/NCI.0b013e3181ac2551. PMID 19638746
- [Background] Dowdy DW, Dinglas V, Mendez-Tellez PA, Bienvenu OJ, Sevransky J, Dennison CR, Shanholtz C, Needham DM. Intensive care unit hypoglycemia predicts depression during early recovery from acute lung injury. Crit Care Med. 2008 Oct;36(10):2726-33. doi: 10.1097/CCM.0b013e31818781f5. PMID 18766087
- [Derived] Al-Dorzi HM, Stapleton RD, Arabi YM. Nutrition priorities in obese critically ill patients. Curr Opin Clin Nutr Metab Care. 2022 Mar 1;25(2):99-109. doi: 10.1097/MCO.0000000000000803. PMID 34930871
- [Derived] Heyland DK, Day A, Clarke GJ, Hough CT, Files DC, Mourtzakis M, Deutz N, Needham DM, Stapleton R. Nutrition and Exercise in Critical Illness Trial (NEXIS Trial): a protocol of a multicentred, randomised controlled trial of combined cycle ergometry and amino acid supplementation commenced early during critical illness. BMJ Open. 2019 Jul 31;9(7):e027893. doi: 10.1136/bmjopen-2018-027893. PMID 31371287